CLINICAL TRIAL: NCT00843921
Title: N-Carbamylglutamate (Carbaglu) In The Treatment Of Hyperammonemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mendel Tuchman (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Mendel Tuchman, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNMC 3694; 1R01HD058567-01 (NIH)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Inborn Errors of Metabolism
Keywords: Hyperammonemia
MeSH Terms: conditions — Metabolism, Inborn Errors; Hyperammonemia | interventions — N-carbamylglutamate; carglumic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carbaglu (Experimental): Investigate whether a 3-day treatment with NCG can improve or restore urea genesis capacity in patients with NAGS, CPSI, or OTC deficiency or PA or MMA using surrogate markers: [13C] label incorporation into urea and plasma levels of ammonia, urea nitrogen (BUN) and amino acids
  Interventions: Drug: N-carbamylglutamate

INTERVENTIONS:
Drug: N-carbamylglutamate — 100 mg/kg/day or 2.2 g/M2/day in 3-4 divided doses for 3 days
  Other Names: Carglumic acid, Carbaglu

SUMMARY:
This study is based on the hypothesis that a new drug N-carbamylglutamate (Carbaglu®) will enhance the ability of the liver to dispose of toxic ammonia which accumulates in several metabolic diseases including urea cycle disorders and organic acid disorders.

DETAILED DESCRIPTION:
Hyperammonemia associated with several rare inherited disorders frequently causes mental retardation, developmental disabilities and death. The overall goal of this study is to investigate the short-term efficacy and safety of the orphan drug, N-Carbamyl-L-glutamate (Carbaglu®, abbreviated as NCG), for the treatment of hyperammonemia in rare inherited disorders: carbamyl phosphate synthetase I (CPSI) deficiency, NAGS deficiency, ornithine transcarbamylase (OTC) deficiency, propionic acidemia (PA) and methylmalonic acidemia (MMA).

The primary aims are:

1. To investigate whether 3-day treatment with NCG can improve or restore ureagenesis capacity in patients with NAGS, CPSI or OTC deficiency using as surrogate markers: [13C] label incorporation into urea and plasma levels of ammonia, urea and glutamine. In addition, to determine whether treatment with NCG in OTC deficiency increases the production of a nitrogen containing intermediate, orotic acid, as a mechanism for eliminating nitrogen in lieu of urea.
2. To investigate whether ureagenesis capacity is deficient in patients with PA and MMA and whether 3-day treatment with NCG can improve or restore ureagenesis capacity in all or some of these patients.
3. To evaluate the safety of short-term (3-day) treatment with NCG in the above patients using clinical and laboratory parameters.

The hypothesis is that ureagenesis capacity as evidenced by [13C] incorporation into urea is deficient in each of these five disorders and that treatment with NCG will improve or restore ureagenesis in patients affected by them. The study will be conducted in the General Clinical Research Centers (GCRC) of the Children's National Medical Center, Washington, D.C. and the Children's Hospital of Philadelphia. Patients (1 day to 70 years of age) with any of the five disorders are eligible for the study. They will all be tested in a short-term trial using surrogate markers (incorporation of [13C] label from Na-acetate into urea, and plasma levels of ammonia, urea and glutamine) before and immediately following 3 days of treatment with NCG. The patients will also be evaluated for short-term safety of NCG using clinical and laboratory parameters. The results of this study will provide important efficacy data, which should help to bring Carbaglu®) to the US market for the benefit of patients with any of these orphan diseases found to be responsive to NCG in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Between 1 day - 70 years of age
2. Viable neonates, neonates with uncertain viability are excluded Diagnosed with one of the following five inborn errors of metabolism: NAGS, CPSI,PA, MMA, or OTC deficiency.
3. Diagnostic requirements:

   * NAGS deficiency - Identification of pathogenic mutation and/or decreased (<20% of control) NAGS enzyme activity in liver
   * CPSI deficiency - decreased (<20% of control) CPSI enzyme activity in liver deficiency of liver CPSI in the presence of normal or substantial activity of OTC (Tuchman et al 1980) and/or molecular confirmation of deleterious mutations (Summary et al 2003).
   * High level of clinical suspicion of NAGS or CPSI deficiency - Failure to meet diagnostic criteria for either NAGS or CPSI deficiency as listed above, but:

     1. Recurrent hyperammonemic episodes (NH3 >70umol/l) with elevated plasma glutamine (>/= 800umol/l)
     2. Urinary orotate levels within normal limits (</= 5 umol/mmol urine creatinine)
     3. Absence of argininosuccinic acid in blood or urine
     4. Low or normal level of citrulline (</=92umol/l) and arginine (</= 179 umol/l) and ornithine (</=159umol/l) within normal limits in blood
   * OTC deficiency- Identification of pathogenic mutation and/or-pedigree analysis consistent with familial hyperammonemia segregating in an x-linked semi-dominant pattern and/or -<20% of control OTC activity in liver and/or -elevated urinary orotate (>20%umol/mmol creatinine) after allopurinol challenge test
   * PA and MMA- diagnostic urine organic acid analysis and confirmation of absence of responsiveness to biotin and vitamin B12 respectively.

Exclusion Criteria:

* Subjects acutely ill on day of the study
* Pregnant females- documentation of a negative pregnancy test within a week prior to testing is required for females 12 years and older, unless having a menstrual period during that week or other circumstances which preclude pregnancy (e.g. hysterectomy, menopause)
* Subjects with hyperammonemia caused by other urea cycle disorders, lysinuric protein intolerance, mitochondrial disorders, congenital lactic academia, fatty acid oxidation defects and primary liver disease
* Subjects requiring a peripherally inserted central catheter (PICC) for blood draws may need to be moderately sedated and are excluded
* Subjects with hemoglobin < 9 g/dl

Ages: 1 Day to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-08; Primary Completion 2018-04-25 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of ureagenesis as determined by 13C enrichment of urea | 3 days of treatment

SECONDARY OUTCOMES:
Plasma ammonia concentration | 3 days
Plasma amino acid levels | 3 days
Urine Orotic Acid | 3 days
  Only in patients with OTC deficiency
Blood Urea Nitrogen (BUN) | 3 days
Routine safety laboratory tests (CBC, LFTs, Creatinine) | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Mendel Tuchman, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with that particular participant